CLINICAL TRIAL: NCT04115020
Title: Low Dose Naltrexone for Chronic Pain in Osteoarthritis and Inflammatory Arthritis
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: A pilot study was negative.
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: VA Boston Healthcare System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Paul Asbury Monach,M.D., Lecturer, Staff Physician, Brigham and Women's Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2019P001799
Record Dates: First submitted 2019-10-02; First posted 2019-10-03 (Actual); Last update posted 2020-01-09 (Actual); Status verified 2020-01

CONDITIONS: Osteoarthritis; Arthritis, Rheumatoid; Arthritis, Psoriatic
MeSH Terms: conditions — Osteoarthritis; Arthritis, Rheumatoid; Arthritis, Psoriatic | interventions — Naltrexone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Naltrexone first then placebo (Experimental): Naltrexone for 8 weeks, then placebo for 8 weeks, blinded cross-over design
  Interventions: Drug: Naltrexone; Drug: Placebo
- Placebo first then naltrexone (Experimental): Placebo for 8 weeks, then naltrexone for 8 weeks, blinded cross-over design
  Interventions: Drug: Naltrexone; Drug: Placebo

INTERVENTIONS:
Drug: Naltrexone — Naltrexone 4.5 mg oral suspension
Drug: Placebo — Placebo oral suspension

SUMMARY:
Over 100 million Americans report chronic pain. One of the most common causes of chronic pain is osteoarthritis (OA). OA is attributable to "wear and tear," but reasons for pain are complex. Inflammatory arthritis (IA) includes multiple severe diseases that affect 2-3% of persons and require treatment with immune-suppressive drugs to prevent joint destruction. Pain often persists despite effective treatment. Pain in arthritis results from multiple sources: inflammation, perception of pain in the joint, and interpretation of pain by the brain. Unfortunately, management of pain in arthritis remains a challenge. Low dose naltrexone is a widely used but unproven "alternative" approach to chronic pain. It is attractive for study because it is safe and is proposed to work on all three pathways that contribute to pain. A small but high-quality clinical trial is needed to determine whether to invest in definitive studies.

DETAILED DESCRIPTION:
Chronic pain affects over 100 million Americans, and arthritis is the most common cause. Existing treatments for chronic arthritic pain are only mildly effective, and risks of medications used to treat pain are numerous and continue to be discovered.

Naltrexone is an opioid antagonist that is FDA approved in an oral daily dose of 50 mg to prevent recidivism in alcoholics. At much lower doses of 4 - 4.5 mg daily, however, it has been shown in small, blinded, randomized trials to improve pain in fibromyalgia, gastrointestinal symptoms in Crohn's disease, and quality of life in multiple sclerosis. The only other published data are case reports in complex regional pain syndrome, low back pain, and scleroderma. However, advocacy of low-dose naltrexone (LDN) by internet-based MDs and patients is high, and since LDN can be prescribed off-label, its use greatly exceeds what is justified by evidence. The drug can be prescribed only via compounding pharmacies, so its use costs a patient ~$40/month.

Among the many unproven treatments that are widely used, LDN is of particular interest because results of surveys of patients are particularly impressive, because it is quite safe, and because its benefit is plausible pharmacologically. There is evidence both for modulation of central pain-processing pathways and for down-regulation of inflammatory pathways in microglia. Considering the diversity of conditions proposed to benefit from LDN and the unequivocal need for better approaches to pain relief in chronic conditions, high-quality clinical trials are needed in both inflammatory and non-inflammatory conditions. This small but placebo-controlled study, powered to detect an effect size as small as that seen with NSAIDs or the most beneficial non-pharmacologic approaches, is being conducted as a prerequisite for considering a pivotal trial.

The proposed study is a randomized, double-blinded, cross-over, placebo-controlled trial in adults with osteoarthritis or inflammatory arthritis and persistent pain. Thirty patients will be enrolled for 16 weeks, during which they will receive LDN for 8 weeks and placebo for 8 weeks. Widely accepted patient-reported outcome measures will be used. The co-primary endpoints are reduction in pain severity or pain's interference with function during 8 weeks of LDN compared to 8 weeks placebo, using the Brief Pain Inventory. Other patient-reported data will be used both as secondary outcomes and as covariates in analyzing determinants of response to treatment. Data from this study will be analyzed in combination with data from a study conducted with 30 patients at the VA, to be completed in 2019. A total of 60 patients in the two studies is sufficient to detect benefit similar to what is seen with NSAIDs.

ELIGIBILITY:
Inclusion Criteria:

* One or more of the following chronic conditions: osteoarthritis, rheumatoid arthritis, or non-axial spondyloarthritis
* Average daily pain interference with function (average of the 7 parts of question 9 on the Brief Pain Inventory) rated at least 4 on a scale of 0-10, and no higher than 9
* No change in medication in the past 8 weeks made with the expectation of improving pain
* No plan to start another medication or a non-pharmacologic treatment regimen likely to affect pain during the next 16 weeks
* Age at least 18
* Capable of informed consent, and willingness to comply with study procedures, including receipt of weekly phone calls from the study coordinator

Exclusion Criteria:

* Use of opioids including tramadol, in the past 7 days
* Pregnant, breast feeding, or unwilling to engage in contraceptive practices if sexually active and capable of conceiving
* Schizophrenia, bipolar disorder, or poorly controlled depression or anxiety
* Previous use of low-dose naltrexone for more than 8 weeks or in the past 2 weeks
* Back pain described by the patient as greater in severity than arthritic pain in all peripheral locations
* Significant kidney disease, defined as glomerular filtration rate < 30 ml/min
* Liver cirrhosis. There is no specific screening procedure to exclude cirrhosis.
* Peripheral neuropathy described by the patient as greater in severity than arthritic pain. There is no specific screening procedure.
* Plan to have surgery during the next 16 weeks
* Other qualitative circumstances that the investigator feels would make the patient a poor candidate for this clinical trial, such as an unstable social situation or unreliable transportation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-01 (Estimated); Primary Completion 2020-01-07 (Actual); Study Completion 2020-01-07 (Actual)

PRIMARY OUTCOMES:
Brief Pain Inventory - Pain Interference | 16 weeks
  Average of 7 questions on how much pain has interfered with general function, walking ability, mood, normal work, relations with other people, sleep, and enjoyment of life

SECONDARY OUTCOMES:
Brief Pain Inventory - Pain Severity | 16 weeks
  Average severity of pain in the past 7 days (0-10)
painDETECT | 16 weeks
  Measure of neuropathic pain (0-38)
Brief Fatigue Inventory | 16 weeks
  Questionnaire, severity of fatigue and fatigue's interference with activity (0-10 scales).
PROMIS-29 | 16 weeks
  Questionnaire, survey of health-related quality of life across 8 domains.
Beck Depression Inventory-II | 16 weeks
  Questionnaire measuring severity of depression. Used primarily during screening to exclude enrollment of patients with severe depression, but also as a safety outcome measure during the study.
Clinical Global Impression of Severity (CGI-S) | 16 weeks
  7-point scale of patients' self-reporting of severity during the study.
Clinical Global Impression of Improvement (CGI-I) | 16 weeks
  7-point scale of patients' self-reporting of improvement or worsening during the study
Pressure-pain threshold testing | 16 weeks
  Measurement of minimum pressure needed to cause detectable pain at each knee
DAS-28 | 16 weeks
  Assessment of disease activity in rheumatoid arthritis (only for patients with rheumatoid arthritis)
BASDAI | 16 weeks
  Assessment of disease activity by MD in spondyloarthritis (only for patients with spondyloarthritis)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Monach, MD, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
A de-identified, anonymized dataset containing all the primary study data will be created and shared consistent with institutional policies. This dataset will be included as a supplementary file attached to the published manuscript, which in turn will be available through PubMed Central. In the event that the study has not been published, the dataset will be made available by other means within 3 years of study completion. The publicly available dataset will not include any identifiers, e.g. age will be included but not birthdate
Supporting Information: Study Protocol
Time Frame: Protocol will be uploaded when results are reported.